CLINICAL TRIAL: NCT03661229
Title: Cardiovascular and Respiratory Assessment Using Biometric Signals in a Non-contact Monitoring Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to demonstrate efficacy. The reason for this is that we were unable to get the necessary information from our population of dialysis patient using the mCVI™ non-contact facial tracking cell phone app.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Intelomed, Inc. (Industry)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, Medical Biophysics and Paediatrics, Robert Lindsay Chair of Dialysis Research and Innovation, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112553
Record Dates: First submitted 2018-08-22; First posted 2018-09-07 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: End-stage Renal Disease
Keywords: CVInsight; Hemodialysis; Cardiovascular stress
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Up to 50 patients will be assessed using the CVInsight Monitoring System. Patients will undergo two consecutive hemodialysis (HD) treatments where they will be monitored with the contact and non-contact devices throughout their HD session. The first visit will be on their first HD session of the week (after the weekend - 72 hour inter-dialytic period) and the second visit will be during the patient's second HD session of the week (mid-week - 48 hour inter-dialytic period). This will allow us to see if there is a difference between these two intervals of time.
  Twenty of these patients will have additional monitoring including movement of left ventricle using echocardiography and continuous blood pressure monitoring using a finometer. The first echocardiogram will be done prior to the initiation of HD and the second at peak HD stress, which is 15 minutes before the end of the HD treatment. 20/50 patients will be chosen according to patient treatment schedule and staff schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CVInsight Monitoring (Experimental): Single group arm: All participants receive the same intervention/treatment CVInsight non-contact device and CVInsight contact device application.
  Interventions: Device: CVInsight Monitoring

INTERVENTIONS:
Device: CVInsight Monitoring — All participants (n=50) will receive CVInsight non-contact device and CVInsight contact device application during two of their regularly scheduled dialysis sessions.

SUMMARY:
Patients on hemodialysis treatment experience increased levels of cardiovascular disease. In this study, investigators will be detecting hemodialysis induced circulatory stress using the CVInsight Patient Monitoring & Informatics System - InteloMed. This system consists of the CVInsight non-contact device and the CVInsight contact device that measures a patient's response to dialysis by looking at many physiological parameters such as heart rate, heart rate variability, respiratory rate, and how much oxygen the blood is carrying. Investigators would like to validate the mobile CVInsight non-contact device to the currently used standard CVInsight contact device to provide healthcare providers with a better understanding of its role in early detection of cardiovascular stress induced by hemodialysis.

DETAILED DESCRIPTION:
This observational validation trial involves patients from the prevalent dialysis population in London, Ontario. Investigators intend to validate the mobile CVInsight non-contact device to the standard contact version of this device for assessing hemodialysis induced circulatory stress. The CVInsight Patient Monitoring & Informatics System records a patient's pulse waveform to determine a patient's response to dialysis and alerts to several physiologic changes including pulse strength, pulse rate, pulse irregularity, oxygen saturation, and oxygen saturation variability. The CVInsight contact and non-contact devices will be used for two study visits. The first study visit will be on the patient's first dialysis session of the week (after the weekend - 72 hour inter-dialytic period) and the second study visit will be during the patient's second dialysis session of the week (mid week - 48 hour inter-dialytic period). This will allow investigators to see if there is a difference between these two intervals of time. The investigators will also be using other gold standard methods of validating components of this device including myocardial stunning using the GE Healthcare Vivid q cardiovascular ultrasound system. The echocardiographic ultrasound machine and finometer will be used for two study visits to take place during the patients' regularly scheduled dialysis sessions. The first echocardiogram will be done prior to the initiation of dialysis and the second at peak dialysis stress, which is 15 minutes before the end of the hemodialysis treatment. In addition, the finometer will be used continuously throughout hemodialysis.Validating the mobile CVInsight non-contact device to the CVInsight contact device will allow investigators to observe the degree to which these devices are able to detect hemodialysis induced circulatory stress, which will enable the healthcare provider to detect injury early enough to intervene prior to its occurrence. This is important because hemodialysis and the accompanying stress it induces increases mortality significantly in this population of patients.

This study is investigator initiated and the study will continue until the investigators reach our target sample size.

Each patient will have two study visits. Patients on a Monday, Wednesday, and Friday schedule will have study visits on Monday and Wednesday of the same week and patients on a Tuesday, Thursday, and Saturday schedule will have study visits on Tuesday and Thursday of the same week.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving conventional thrice weekly maintenance HD
* Age ≥18 years
* Able to provide informed consent

Exclusion Criteria:

• Not meeting inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Mobile CVInsight validation against the CVInsight contact device by recording pulse rate trends | Through dialysis session, an average of 4 hours for two separate visits within the same week.
  Validation of the mobile CVInsight with pulse rate from the CVInsight contact device
Mobile CVInsight validation against the CVInsight contact device by recording pulse strength | Through dialysis session, an average of 4 hours for two separate visits within the same week.
  Validation of the mobile CVInsight with pulse strength (derived from a photoelectric plethysmograph waveform) from the CVInsight contact device
Mobile CVInsight validation against the CVInsight contact device by recording pulse irregularity | Through dialysis session, an average of 4 hours for two separate visits within the same week.
  Validation of the mobile CVInsight with pulse irregularity (derived from the pulse wave signal) from the CVInsight contact device
Mobile CVInsight validation against the CVInsight contact device by recording oxygen saturation | Through dialysis session, an average of 4 hours for two separate visits within the same week.
  Validation of the mobile CVInsight with the percentage of oxygen carried in blood from the CVInsight contact device
Mobile CVInsight validation against the CVInsight contact device by recording oxygen saturation variability | Through dialysis session, an average of 4 hours for two separate visits within the same week.
  Validation of the mobile CVInsight with the oxygen saturation variability (derived from the oximeter signal) from the CVInsight contact device

SECONDARY OUTCOMES:
Early detection of hemodialysis-induced circulatory stress using the CVInsight System | Through dialysis session, an average of 4 hours for two separate visits within the same week.
  The secondary outcome will be assessment of the contact and non-contact CVInsight devices on hemodialysis induced circulatory stress
Early detection of hemodialysis-induced circulatory stress using the finometer | Through dialysis session, an average of 4 hours for two separate visits within the same week.
  The secondary outcome will be assessment of the finometer on hemodialysis induced circulatory stress
Early detection of hemodialysis-induced circulatory stress using echocardiography | Before the dialysis session and 15 minutes prior to the end of the dialysis session for two separate visits within the same week.
  The secondary outcome will be assessment of echocardiography on hemodialysis induced circulatory stress

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McIntyre, MBBS DM, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada